CLINICAL TRIAL: NCT04300296
Title: A Proof of Concept Study to Evaluate the Efficacy, Safety and Tolerability of Secukinumab 300 mg Over 32 Weeks in Adult Patients With Biopsy-proven Forms of Lichen Planus Not Adequately Controlled With Topical Therapies - PRELUDE
Brief Title: PoC Study to Evaluate the Efficacy and Safety of Secukinumab 300 mg in Patients With Lichen Planus
Acronym: PRELUDE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457S12201; 2019-003588-24 (EudraCT Number)
Record Dates: First submitted 2020-01-08; First posted 2020-03-09 (Actual); Results first posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-07

CONDITIONS: Lichen Planus: Cutaneous Lichen Planus, Mucosal Lichen Planus and Lichen Planopilaris
Keywords: Lichen planus; CLP; MLP; LPP
MeSH Terms: conditions — Lichen Planus | interventions — secukinumab

STUDY DESIGN:
Intervention Model Description: PoC study, 32-week, multicenter, randomized, double-blind, placebo-controlled, parallel-group trial assessing the efficacy and safety of secukinumab 300 mg in two different dosing regimens in 108 patients with biopsy-proven forms of lichen planus.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Cutaneous lichen planus secukinumab 300mg Q4W (Experimental): Secukinumab 300 mg every 4 weeks provided in pre-filled syringe in cutaneous lichen planus patients
  Interventions: Drug: secukinumab 300 mg Q4W
- Cutaneous lichen planus placebo (Placebo Comparator): Placebo in 1ml PFS in cutaneous lichen patients
  Interventions: Other: Placebo
- Mucosal lichen planus secukinumab 300 mg Q4W (Experimental): Secukinumab 300 mg every 4 weeks provided in pre-filled syringe in mucosal lichen planus patients.
  Interventions: Drug: secukinumab 300 mg Q4W
- Mucosal lichen planus placebo (Placebo Comparator): Placebo 1 ml PFS in mucosal lichen planus patients
  Interventions: Other: Placebo
- Lichen planopilaris secukinumab 300 mg Q4W (Experimental): Secukinumab 300 mg every 4weeks provided in pre-filled syringe in lichen planopilaris patients.
  Interventions: Drug: secukinumab 300 mg Q4W
- Lichen planopilaris placebo (Placebo Comparator): Placebo in 1ml PFS in lichen planopilaris patients
  Interventions: Other: Placebo
- Cutaneous lichen planus placebo to secukinumab 300 mg Q2W (Experimental): Non responder patients on placebo in TP 1 received secukinumab 300 mg Q2W in TP 2
  Interventions: Drug: secukinumab 300 mg Q2W
- Mucosal lichen planus placebo to secukinumab 300 mg Q2W (Experimental): Non responder patients on placebo in TP 1 received secukinumab 300 mg Q2W in TP 2
  Interventions: Drug: secukinumab 300 mg Q2W
- Lichen planopilaris placebo to secukinumab 300 mg Q2W (Experimental): Non responder patients on placebo in TP 1 received secukinumab 300 mg Q2W in TP 2
  Interventions: Drug: secukinumab 300 mg Q2W

INTERVENTIONS:
Drug: secukinumab 300 mg Q4W — secukinumab 300 mg administered every four weeks (Q4W) via a pre-filled syringe.
  Other Names: AIN457
  Arms: Cutaneous lichen planus secukinumab 300mg Q4W; Lichen planopilaris secukinumab 300 mg Q4W; Mucosal lichen planus secukinumab 300 mg Q4W
Drug: secukinumab 300 mg Q2W — secukinumab 300 mg administered every two weeks (Q2W) via a pre-filled syringe.
  Other Names: AIN457
  Arms: Cutaneous lichen planus placebo to secukinumab 300 mg Q2W; Lichen planopilaris placebo to secukinumab 300 mg Q2W; Mucosal lichen planus placebo to secukinumab 300 mg Q2W
Other: Placebo — Matching placebo administered via a pre-filled syringe
  Arms: Cutaneous lichen planus placebo; Lichen planopilaris placebo; Mucosal lichen planus placebo

SUMMARY:
The primary purpose of the proof of concept study is to elucidate the efficacy of secukinumab in the treatment of adult patients with biopsy-proven lichen planus not adequately controlled by topical therapies, and to assess the safety and tolerability over 32 weeks.

DETAILED DESCRIPTION:
This was a 32-week, multicenter, randomized, double-blind, placebo-controlled, parallel-group trial which assessed the efficacy and safety of secukinumab 300 mg in two different dosing regimens: every 4 weeks (Q4W) and every 2 weeks (Q2W) in approximately 111 patients with biopsy-proven forms of lichen planus.

There was a screening period (up to 4 weeks prior to baseline), a treatment period 1 (baseline to Week 16), a treatment period 2 (Week 16 to Week 32) and a follow-up period (8 weeks after Week 32).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any assessment is performed.
2. Female and male patients ≥ 18 years of age.
3. Subjects must have biopsy-confirmed forms of cutaneous lichen planus (CLP), mucosal lichen planus (MLP), or active lichen planopilaris (LPP) eligible for systemic therapy based on the following criteria:

   * rated IGA of ≥ 3 (moderate or severe) AND
   * inadequate response to topical corticosteroids of high-ultrahigh potency in the opinion of the investigator.
4. If using any of the allowed topical treatments on the affected areas, the dose and application frequency should remain stable for 2 weeks prior to randomization and until Week 16.

Exclusion Criteria:

1. Clinical history suspicious for lichenoid drug eruption.
2. Lichen planus pigmentosus.
3. Clinical picture or history suspicious of paraneoplastic mucosal lichen planus.
4. Subjects whose lichen planus is a predominantly bullous variant.
5. Mucosal LP of the oral cavity or gastrointestinal involvement requiring the patient to use parenteral nutrition or feeding tube.
6. Clinical picture of scarring alopecia without active inflammation.
7. Clinical picture of burnt-out cicatricial alopecia (alopecia of Brocque).
8. Patients diagnosed with frontal fibrosing alopecia (FFA) without active patches of LPP
9. Clinical picture of LPP in patients who have already failed 3 or more systemic immunosuppressive or immunomodulatory agents (e.g. systemic steroids, hydroxychloroquine, cyclosporine, methotrexate and mycophenolate mofetil).
10. Currently enrolled in any other clinical trial involving any investigational agent or device.
11. Previous exposure to any other biologic drug directly targeting IL-17A or IL-17RA (e.g. secukinumab, ixekizumab or brodalumab) or IL-23/p19 (e.g. tildrakizumab, guselkumab, risankizumab).
12. Diagnosis of active infectious diseases of the skin, scalp or mucosa (for example bacterial, viral or fungal infections of the mouth) that may interfere with the assessment of the study disease or require treatment with prohibited medications.
13. Diagnosis of active inflammatory diseases of the skin, scalp or mucosa other than lichen planus that may interfere with the assessment of the study disease or require treatment with prohibited medications.
14. Presence of any other skin condition that may affect the evaluations of the study disease.
15. Underlying conditions (including, but not limited to metabolic, hematologic, renal, hepatic, pulmonary, neurologic, endocrine, cardiac, infectious or gastrointestinal) and/or presence of laboratory abnormalities which in the opinion of the investigator significantly immunocompromises the subject and/or places the subject at unacceptable risk for receiving an immunomodulatory therapy.
16. Current, severe, progressive or uncontrolled diseases that render the patient unsuitable for the trial, including any medical or psychiatric condition that, in the Investigator's opinion, would preclude the participant from adhering to the protocol or completing the study per protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2021-11-16 (Actual); Study Completion 2022-05-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (35):
- United States (15):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Thousand Oaks, California
  - Novartis Investigative Site, Cromwell, Connecticut
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Snellville, Georgia
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, East Windsor, New Jersey
  - Novartis Investigative Site, Forest Hills, New York
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Pflugerville, Texas
- France (9):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Chambray-lès-Tours
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Toulouse
- Germany (11):
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bramsche
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Würzburg

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Mahon-Smith A, Skingley G, Ayala-Nunes L, Batish A, Sharp R, Naujoks C, Schruf E, Compagno N, Moreno SG. Evaluating the Appropriateness of Existing Health-Related Quality of Life Measures in Lichen Planus. Dermatol Ther (Heidelb). 2023 Nov;13(11):2817-2837. doi: 10.1007/s13555-023-00990-4. Epub 2023 Oct 5. PMID 37794275
- [Derived] Mahon-Smith A, Clifford M, Batish A, Sharp R, Panter C, Naujoks C, Schruf E, Compagno N, Moreno SG. Patient Experience of Lichen Planus: A Qualitative Exploration of Signs, Symptoms, and Health-Related Quality of Life Impacts. Dermatol Ther (Heidelb). 2023 Sep;13(9):2001-2017. doi: 10.1007/s13555-023-00968-2. Epub 2023 Jul 28. PMID 37505393
- [Derived] Miteva M, Nadji M, Billero V, LaSenna C, Nattkemper L, Romanelli P. IL-17 Expression in the Perifollicular Fibrosis in Biopsies From Lichen Planopilaris. Am J Dermatopathol. 2022 Dec 1;44(12):874-878. doi: 10.1097/DAD.0000000000002316. Epub 2022 Sep 27. PMID 36197049

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 163 subjects (3 cohorts) were screened and 111 were randomized. Subjects in the AIN457 300 mg Q4W group in TP1 continued on AIN457 300mg Q4W in TP2. Subjects in the Placebo group in TP1 received AIN457 300mg Q2W in TP2. Patients in the Placebo group with spontaneous remission at Week 16 entered the Follow-up period.
Groups:
- AIN457 300 mg Q4W - TP 1 and TP 2 - CLP Cohort; AIN457 300 mg Q4W - TP 1 and TP 2 - MLP Cohort; AIN457 300 mg Q4W - TP 1 and TP 2 - LPP Cohort: AIN457 300 mg every 4 weeks administered via a pre-filled syringe. Participants on AIN457 in TP 1 for 16 weeks continued AIN457 in TP 2 for 16 weeks.
- Placebo in TP1 to AIN457 300 mg Q2W - TP 2 - CLP Cohort; Placebo in TP1 to AIN457 300 mg Q2W - TP 2 - MLP Cohort; Placebo in TP1 to AIN457 300 mg Q2W - TP 2 - LPP Cohort: Placebo in TP1. Placebo non-responders during TP 1 received AIN457 300 mg every 2 weeks from Week 16 to Week 32 in TP 2 via a pre-filled syringe
Period: Treatment Period 1: Baseline to 16 Weeks
Arm/Group | AIN457 300 mg Q4W - TP 1 and TP 2 - CLP Cohort | Placebo in TP1 to AIN457 300 mg Q2W - TP 2 - CLP Cohort | AIN457 300 mg Q4W - TP 1 and TP 2 - MLP Cohort | Placebo in TP1 to AIN457 300 mg Q2W - TP 2 - MLP Cohort | AIN457 300 mg Q4W - TP 1 and TP 2 - LPP Cohort | Placebo in TP1 to AIN457 300 mg Q2W - TP 2 - LPP Cohort
Started | 25 | 12 | 24 | 13 | 24 | 13
Placebo Responder | 0 | 1 | 0 | 1 | 0 | 0
Completed | 23 | 10 | 24 | 13 | 23 | 12
Not Completed | 2 | 2 | 0 | 0 | 1 | 1
Not completed — Progressive disease | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Subject/guardian decision | 1 | 2 | 0 | 0 | 0 | 1
Period: Treatment Period 2: 16 to 32 Weeks
Arm/Group | AIN457 300 mg Q4W - TP 1 and TP 2 - CLP Cohort | Placebo in TP1 to AIN457 300 mg Q2W - TP 2 - CLP Cohort | AIN457 300 mg Q4W - TP 1 and TP 2 - MLP Cohort | Placebo in TP1 to AIN457 300 mg Q2W - TP 2 - MLP Cohort | AIN457 300 mg Q4W - TP 1 and TP 2 - LPP Cohort | Placebo in TP1 to AIN457 300 mg Q2W - TP 2 - LPP Cohort
Started | 22 | 8 | 23 | 11 | 23 | 12
Completed | 17 | 7 | 19 | 10 | 17 | 12
Not Completed | 5 | 1 | 4 | 1 | 6 | 0
Not completed — Adverse Event | 1 | 0 | 2 | 0 | 1 | 0
Not completed — Progressive disease | 2 | 0 | 1 | 0 | 2 | 0
Not completed — Protocol deviation | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Subject/guardian decision | 2 | 0 | 1 | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- AIN457 300 mg Q4W - TP 1 - CLP Cohort; AIN457 300 mg Q4W - TP 1 - MLP Cohort: AIN457 300 mg every 4 weeks up to 16 weeks administered via a pre-filled syringe
- Placebo - TP 1 - CLP Cohort; Placebo - TP 1 - MLP Cohort; Placebo - TP 1 - LPP Cohort: Matching placebo administered every 4 weeks up to 16 weeks via a pre-filled syringe
- AIN457 300 mg Q4W - TP 1 - LPP Cohort: AIN457457 300 mg every 4 weeks up to 16 weeks administered via a pre-filled syringe
- Total: Total of all reporting groups
Arm/Group | AIN457 300 mg Q4W - TP 1 - CLP Cohort | Placebo - TP 1 - CLP Cohort | AIN457 300 mg Q4W - TP 1 - MLP Cohort | Placebo - TP 1 - MLP Cohort | AIN457 300 mg Q4W - TP 1 - LPP Cohort | Placebo - TP 1 - LPP Cohort | Total
Number analyzed (Participants) | 25 | 12 | 24 | 13 | 24 | 13 | 111
Age, Customized [Number; unit: Participants]
  18 to <65 years | 22 | 9 | 14 | 8 | 19 | 12 | 84
  > or = 65 years | 3 | 3 | 10 | 5 | 5 | 1 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 8 | 14 | 12 | 20 | 10 | 79
  Male | 10 | 4 | 10 | 1 | 4 | 3 | 32
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian (Indian) | 0 | 0 | 2 | 0 | 0 | 0 | 2
  Black or African American | 6 | 4 | 2 | 1 | 1 | 0 | 14
  White | 19 | 8 | 19 | 12 | 23 | 13 | 94
  White, American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 0 | 1
Baseline of Investigator's Global Assessment (IGA) [Count of Participants; unit: Participants] — The IGA provides a harmonized, 5-point grading system to assess disease severity for subjects of all 3 subtypes entering the study. The predominant subtype alone defined the IGA score of the subject and was collected separately for concomitant subtypes, if present (0=clear, 1=minimal, 2=mild, 3=moderate, 4=severe).
  Participants
    0=Clear | 0 | 0 | 0 | 0 | 0 | 0 | 0
    1=Minimal | 1 | 0 | 0 | 0 | 0 | 0 | 1
    2=Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0
    3=Moderate | 16 | 9 | 22 | 8 | 17 | 10 | 82
    4=Severe | 8 | 3 | 2 | 5 | 7 | 3 | 28

OUTCOME MEASURES:

1. Primary Outcome: Response Rate of Investigator Global Assessment (IGA) Score of 2 or Lower at Week 16 for CLP, MLP and LPP
Description: Number of treatment responders at week 16, where response is defined as an Investigator's Global Assessment (IGA) score of 2 or lower at Week 16. IGA is measured on a scale from 0 - 4 with 0 = Clear, 1 = Minimal; 2 = Mild; 3 = Moderate; and 4 = Severe with 0 being best score and 4 being worst score. CLP=Cutaneous lichen planus, MLP=Mucosal lichen planus, LPP=Lichen planopilaris. Posterior median and 95% credible interval (instead of 95% confidence interval) were derived using Bayesian method based on beta-binomial model.
Time Frame: Baseline up to week 16
Population: Full analysis set of participants with a baseline IGA score >= 3 were included
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | AIN457 300 mg Q4W - TP 1 - CLP Cohort | Placebo - TP 1 - CLP Cohort | AIN457 300 mg Q4W - TP 1 - MLP Cohort | Placebo - TP 1 - MLP Cohort | AIN457 300 mg Q4W - TP 1 - LPP Cohort | Placebo - TP 1 - LPP Cohort
Number analyzed (Participants) | 25 | 12 | 24 | 13 | 24 | 13
percentage of participants | 44.0 [25.8 to 63.32] | 58.2 [31.0 to 82.6] | 37.5 [20.3 to 57.2] | 23.1 [6.5 to 49.2] | 37.6 [20.2 to 57.3] | 30.9 [10.8 to 57.6]
Statistical Analysis 1: Comparison: AIN457 300 mg Q4W - TP 1 - CLP Cohort vs Placebo - TP 1 - CLP Cohort; Test type: Other; Posterior median difference = -13.9, 95% CI 2-sided [-44.8 to 19.3] — Bayesian model to obtain the posterior distribution of the treatment difference between AIN457 and placebo
Statistical Analysis 2: Comparison: AIN457 300 mg Q4W - TP 1 - MLP Cohort vs Placebo - TP 1 - MLP Cohort; Test type: Other; Posterior median difference = 14.1, 95% CI 2-sided [-17.0 to 40.7] — Bayesian model to obtain the posterior distribution of the treatment difference between AIN457 and placebo
Statistical Analysis 3: Comparison: AIN457 300 mg Q4W - TP 1 - LPP Cohort vs Placebo - TP 1 - LPP Cohort; Test type: Other; Posterior median difference = 6.5, 95% CI 2-sided [-25.4 to 35.4] — Bayesian model to obtain the posterior distribution of the treatment difference between AIN457 and placebo

2. Secondary Outcome: Number (%) of Subjects With IGA ≤ 2 Response, IGA ≥2 Points Improvement Response, and IGA 0 or 1 Response by Visit - CLP Cohort (BOCF)- Entire Treatment Period (FAS)
Description: Number of subjects with IGA of 2 or lower, improvement in the IGA score of at least 2 points, or IGA score of 0/1. IGA is measured on a scale from 0-4 with 0=Clear, 1=minimal, 2=mild, 3=moderate, and 4=severe with 0 being best score and 4 being worst score.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, 28, and 32
Population: Full analysis set. Patients who were included in FAS for TP1 were included in FAS for TP2 except that the placebo patients in spontaneous remission at Week 16 were excluded from Placebo- AIN457 300 mg Q2W TP2 group. Patients who discontinued study treatment before week 32 were imputed using baseline observation carried forward. Missing values not related to treatment discontinuation were analyzed as observed.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo to AIN457 300 mg Q2W - TP 2 - CLP Cohort: Placebo non-responders during TP 1 received AIN457 300 mg every 2 weeks from Week 16 to Week 32 in TP 2 via a pre-filled syringe.
Arm/Group | AIN457 300 mg Q4W - TP 1 and TP 2 - CLP Cohort | Placebo - TP 1 - CLP Cohort | Placebo to AIN457 300 mg Q2W - TP 2 - CLP Cohort
Number analyzed (Participants) | 25 | 12 | 10
Participants
  Week 2 IGA <=2 n=25,12,0: number analyzed (Participants) | 25 | 12 | 0
  Week 2 IGA <=2 n=25,12,0 | 5 | 1 |
  Week 2 IGA improvement >=2 n=25,12,0: number analyzed (Participants) | 25 | 12 | 0
  Week 2 IGA improvement >=2 n=25,12,0 | 2 | 0 |
  Week 2 IGA 0/1 n=25,12,0: number analyzed (Participants) | 25 | 12 | 0
  Week 2 IGA 0/1 n=25,12,0 | 2 | 0 |
  Week 4 IGA <=2 n=24,11,0: number analyzed (Participants) | 24 | 11 | 0
  Week 4 IGA <=2 n=24,11,0 | 9 | 2 |
  Week 4 IGA improvement. >=2 n=24,11,0: number analyzed (Participants) | 24 | 11 | 0
  Week 4 IGA improvement. >=2 n=24,11,0 | 3 | 0 |
  Week 4 IGA 0/1 n=24,11,0: number analyzed (Participants) | 24 | 11 | 0
  Week 4 IGA 0/1 n=24,11,0 | 2 | 0 |
  Week 8 IGA <=2 n=25,11,0: number analyzed (Participants) | 25 | 11 | 0
  Week 8 IGA <=2 n=25,11,0 | 10 | 3 |
  Week 8 IGA improvement. >=2 n=25,11,0: number analyzed (Participants) | 25 | 11 | 0
  Week 8 IGA improvement. >=2 n=25,11,0 | 4 | 1 |
  Week 8 IGA 0/1 n=25,11,0: number analyzed (Participants) | 25 | 11 | 0
  Week 8 IGA 0/1 n=25,11,0 | 3 | 1 |
  Week 12 IGA <=2 n=25,12,0: number analyzed (Participants) | 25 | 12 | 0
  Week 12 IGA <=2 n=25,12,0 | 10 | 4 |
  Week 12 IGA improvement. >=2 n=25,12,0: number analyzed (Participants) | 25 | 12 | 0
  Week 12 IGA improvement. >=2 n=25,12,0 | 3 | 2 |
  Week 12 IGA 0/1 n=25,12,0: number analyzed (Participants) | 25 | 12 | 0
  Week 12 IGA 0/1 n=25,12,0 | 4 | 1 |
  Week16 IGA <=2 n=25,12,10 | 11 | 7 | 5
  Week 16 IGA improvement. >=2 n=25,12,10 | 4 | 3 | 1
  Week 16 IGA 0/1 n=25,12,10 | 4 | 2 | 0
  Week 20 IGA <=2 n=24,0,10: number analyzed (Participants) | 24 | 0 | 10
  Week 20 IGA <=2 n=24,0,10 | 11 |  | 1
  Week 20 IGA improvement. >=2 n=24,0,10: number analyzed (Participants) | 24 | 0 | 10
  Week 20 IGA improvement. >=2 n=24,0,10 | 5 |  | 1
  Week 20 IGA 0/1 n=24,0,10: number analyzed (Participants) | 24 | 0 | 10
  Week 20 IGA 0/1 n=24,0,10 | 5 |  | 1
  Week 24 IGA <=2 n=25,0,10: number analyzed (Participants) | 25 | 0 | 10
  Week 24 IGA <=2 n=25,0,10 | 14 |  | 3
  Week 24 IGA improvement. >=2 n=25,0,10: number analyzed (Participants) | 25 | 0 | 10
  Week 24 IGA improvement. >=2 n=25,0,10 | 10 |  | 2
  Week 24 IGA 0/1 n=25,0,10: number analyzed (Participants) | 25 | 0 | 10
  Week 24 IGA 0/1 n=25,0,10 | 10 |  | 1
  Week 28 IGA <=2 n=23,0,10: number analyzed (Participants) | 23 | 0 | 10
  Week 28 IGA <=2 n=23,0,10 | 12 |  | 4
  Week 28 IGA improvement. >=2 n=23,0,10: number analyzed (Participants) | 23 | 0 | 10
  Week 28 IGA improvement. >=2 n=23,0,10 | 7 |  | 1
  Week 28 IGA 0/1 n=23,0,10: number analyzed (Participants) | 23 | 0 | 10
  Week 28 IGA 0/1 n=23,0,10 | 6 |  | 1
  Week 32 IGA <=2 n=24,0,9: number analyzed (Participants) | 24 | 0 | 9
  Week 32 IGA <=2 n=24,0,9 | 9 |  | 2
  Week 32 IGA improvement. >=2 n=24,0,9: number analyzed (Participants) | 24 | 0 | 9
  Week 32 IGA improvement. >=2 n=24,0,9 | 7 |  | 2
  Week 32 IGA 0/1 n=24,0,9: number analyzed (Participants) | 24 | 0 | 9
  Week 32 IGA 0/1 n=24,0,9 | 6 |  | 1

3. Secondary Outcome: Number (%) of Subjects With IGA ≤ 2 Response, IGA ≥2 Points Improvement Response, and IGA 0 or 1 Response by Visit - MLP Cohort (BOCF)- Entire Treatment Period (FAS)
Description: Number of subjects with IGA of 2 of lower, improvement in the IGA score of at least 2 points, or IGA score of 0/1. IGA is measured on a scale from 0-4 with 0=Clear, 1=minimal, 2=mild, 3=moderate, and 4=severe with 0 being best score and 4 being worst score.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, 28, and 32
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Placebo to AIN457 300 mg Q2W TP 2 - MLP Cohort: Placebo non-responders during TP 1 received AIN457 300 mg every 2 weeks from Week 16 to Week 32 in TP 2 via a pre-filled syringe.
Arm/Group | AIN457 300 mg Q4W - TP 1 and TP 2 - MLP Cohort | Placebo - TP 1 - MLP Cohort | Placebo to AIN457 300 mg Q2W TP 2 - MLP Cohort
Number analyzed (Participants) | 24 | 13 | 11
Participants
  Week 2 IGA <=2 n=24,12,0: number analyzed (Participants) | 24 | 12 | 0
  Week 2 IGA <=2 n=24,12,0 | 5 | 3 |
  Week 2 IGA improvement >=2 n=24,12,0: number analyzed (Participants) | 24 | 12 | 0
  Week 2 IGA improvement >=2 n=24,12,0 | 1 | 1 |
  Week 2 IGA 0/1 n=24,12,0: number analyzed (Participants) | 24 | 12 | 0
  Week 2 IGA 0/1 n=24,12,0 | 1 | 1 |
  Week 4 IGA <=2 n=24,13,0: number analyzed (Participants) | 24 | 13 | 0
  Week 4 IGA <=2 n=24,13,0 | 4 | 2 |
  Week 4 IGA improvement. >=2 n=24,13,0: number analyzed (Participants) | 24 | 13 | 0
  Week 4 IGA improvement. >=2 n=24,13,0 | 1 | 1 |
  Week 4 IGA 0/1 n=24,13,0: number analyzed (Participants) | 24 | 13 | 0
  Week 4 IGA 0/1 n=24,13,0 | 1 | 1 |
  Week 8 IGA <=2 n=24,13,0: number analyzed (Participants) | 24 | 13 | 0
  Week 8 IGA <=2 n=24,13,0 | 5 | 3 |
  Week 8 IGA improvement. >=2 n=24,13,0: number analyzed (Participants) | 24 | 13 | 0
  Week 8 IGA improvement. >=2 n=24,13,0 | 0 | 2 |
  Week 8 IGA 0/1 n=24,13,0: number analyzed (Participants) | 24 | 13 | 0
  Week 8 IGA 0/1 n=24,13,0 | 0 | 1 |
  Week 12 IGA <=2 n=24,13,0: number analyzed (Participants) | 24 | 13 | 0
  Week 12 IGA <=2 n=24,13,0 | 5 | 4 |
  Week 12 IGA improvement. >=2 n=24,13,0: number analyzed (Participants) | 24 | 13 | 0
  Week 12 IGA improvement. >=2 n=24,13,0 | 5 | 4 |
  Week 12 IGA 0/1 n=24,13,0: number analyzed (Participants) | 24 | 13 | 0
  Week 12 IGA 0/1 n=24,13,0 | 4 | 2 |
  Week16 IGA <=2 n=24,13,11 | 9 | 3 | 1
  Week 16 IGA improvement. >=2 n=24,13,11 | 5 | 3 | 1
  Week 16 IGA 0/1 n=24,13,11 | 4 | 2 | 0
  Week 20 IGA <=2 n=24,0,11: number analyzed (Participants) | 24 | 0 | 11
  Week 20 IGA <=2 n=24,0,11 | 10 |  | 3
  Week 20 IGA improvement. >=2 n=24,0,11: number analyzed (Participants) | 24 | 0 | 11
  Week 20 IGA improvement. >=2 n=24,0,11 | 5 |  | 2
  Week 20 IGA 0/1 n=24,0,11: number analyzed (Participants) | 24 | 0 | 11
  Week 20 IGA 0/1 n=24,0,11 | 5 |  | 1
  Week 24 IGA <=2 n=24,0,10: number analyzed (Participants) | 24 | 0 | 10
  Week 24 IGA <=2 n=24,0,10 | 10 |  | 4
  Week 24 IGA improvement. >=2 n=24,0,10: number analyzed (Participants) | 24 | 0 | 10
  Week 24 IGA improvement. >=2 n=24,0,10 | 3 |  | 2
  Week 24 IGA 0/1 n=24,0,10: number analyzed (Participants) | 24 | 0 | 10
  Week 24 IGA 0/1 n=24,0,10 | 3 |  | 0
  Week 28 IGA <=2 n=23,0,11: number analyzed (Participants) | 23 | 0 | 11
  Week 28 IGA <=2 n=23,0,11 | 7 |  | 4
  Week 28 IGA improvement. >=2 n=23,0,11: number analyzed (Participants) | 23 | 0 | 11
  Week 28 IGA improvement. >=2 n=23,0,11 | 1 |  | 3
  Week 28 IGA 0/1 n=23,0,11: number analyzed (Participants) | 23 | 0 | 11
  Week 28 IGA 0/1 n=23,0,11 | 1 |  | 0
  Week 32 IGA <=2 n=23,0,10: number analyzed (Participants) | 23 | 0 | 10
  Week 32 IGA <=2 n=23,0,10 | 9 |  | 2
  Week 32 IGA improvement. >=2 n=23,0,10: number analyzed (Participants) | 23 | 0 | 10
  Week 32 IGA improvement. >=2 n=23,0,10 | 2 |  | 1
  Week 32 IGA 0/1 n=23,0,10: number analyzed (Participants) | 23 | 0 | 10
  Week 32 IGA 0/1 n=23,0,10 | 2 |  | 0

4. Secondary Outcome: Number (%) of Subjects With IGA ≤ 2 Response, IGA ≥2 Points Improvement Response, and IGA 0 or 1 Response by Visit - LPP Cohort (BOCF)- Entire Treatment Period (FAS)
Description: as for outcome 2
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, 28, and 32
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Placebo to AIN457 300 mg Q2W - TP 2- LPP Cohort: Participants on placebo during Treatment 1 received AIN457 300 mg every 2 weeks administered via a pre-filled syringe
Arm/Group | AIN457 300 mg Q4W - TP 1 and TP 2 - LPP Cohort | Placebo - TP 1 - LPP Cohort | Placebo to AIN457 300 mg Q2W - TP 2- LPP Cohort
Number analyzed (Participants) | 24 | 13 | 13
Participants
  Week 2 IGA <=2 n=24,13,0: number analyzed (Participants) | 24 | 13 | 0
  Week 2 IGA <=2 n=24,13,0 | 4 | 1 |
  Week 2 IGA improvement >=2 n=24,13,0: number analyzed (Participants) | 24 | 13 | 0
  Week 2 IGA improvement >=2 n=24,13,0 | 1 | 0 |
  Week 2 IGA 0/1 n=24,13,0: number analyzed (Participants) | 24 | 13 | 0
  Week 2 IGA 0/1 n=24,13,0 | 1 | 0 |
  Week 4 IGA <=2 n=24,13,0: number analyzed (Participants) | 24 | 13 | 0
  Week 4 IGA <=2 n=24,13,0 | 9 | 2 |
  Week 4 IGA improvement. >=2 n=24,13,0: number analyzed (Participants) | 24 | 13 | 0
  Week 4 IGA improvement. >=2 n=24,13,0 | 2 | 1 |
  Week 4 IGA 0/1 n=24,13,0: number analyzed (Participants) | 24 | 13 | 0
  Week 4 IGA 0/1 n=24,13,0 | 2 | 1 |
  Week 8 IGA <=2 n=24,13,0: number analyzed (Participants) | 24 | 13 | 0
  Week 8 IGA <=2 n=24,13,0 | 8 | 3 |
  Week 8 IGA improvement. >=2 n=24,13,0: number analyzed (Participants) | 24 | 13 | 0
  Week 8 IGA improvement. >=2 n=24,13,0 | 3 | 1 |
  Week 8 IGA 0/1 n=24,13,0: number analyzed (Participants) | 24 | 13 | 0
  Week 8 IGA 0/1 n=24,13,0 | 3 | 1 |
  Week 12 IGA <=2 n=24,13,0: number analyzed (Participants) | 24 | 13 | 0
  Week 12 IGA <=2 n=24,13,0 | 8 | 4 |
  Week 12 IGA improvement. >=2 n=24,13,0: number analyzed (Participants) | 24 | 13 | 0
  Week 12 IGA improvement. >=2 n=24,13,0 | 3 | 2 |
  Week 12 IGA 0/1 n=24,13,0: number analyzed (Participants) | 24 | 13 | 0
  Week 12 IGA 0/1 n=24,13,0 | 2 | 2 |
  Week16 IGA <=2 n=24,13,13 | 9 | 4 | 4
  Week 16 IGA improvement. >=2 n=24,13,13 | 3 | 0 | 0
  Week 16 IGA 0/1 n=24,13,13 | 2 | 0 | 0
  Week 20 IGA <=2 n=24,0,13: number analyzed (Participants) | 24 | 0 | 13
  Week 20 IGA <=2 n=24,0,13 | 10 |  | 6
  Week 20 IGA improvement. >=2 n=24,0,13: number analyzed (Participants) | 24 | 0 | 13
  Week 20 IGA improvement. >=2 n=24,0,13 | 6 |  | 1
  Week 20 IGA 0/1 n=24,0,13: number analyzed (Participants) | 24 | 0 | 13
  Week 20 IGA 0/1 n=24,0,13 | 4 |  | 0
  Week 24 IGA <=2 n=23,0,13: number analyzed (Participants) | 23 | 0 | 13
  Week 24 IGA <=2 n=23,0,13 | 10 |  | 8
  Week 24 IGA improvement. >=2 n=23,0,13: number analyzed (Participants) | 23 | 0 | 13
  Week 24 IGA improvement. >=2 n=23,0,13 | 7 |  | 3
  Week 24 IGA 0/1 n=23,0,13: number analyzed (Participants) | 23 | 0 | 13
  Week 24 IGA 0/1 n=23,0,13 | 6 |  | 2
  Week 28 IGA <=2 n=24,0,13: number analyzed (Participants) | 24 | 0 | 13
  Week 28 IGA <=2 n=24,0,13 | 10 |  | 9
  Week 28 IGA improvement. >=2 n=24,0,13: number analyzed (Participants) | 24 | 0 | 13
  Week 28 IGA improvement. >=2 n=24,0,13 | 6 |  | 4
  Week 28 IGA 0/1 n=24,0,13: number analyzed (Participants) | 24 | 0 | 13
  Week 28 IGA 0/1 n=24,0,13 | 5 |  | 3
  Week 32 IGA <=2 n==24,0,11: number analyzed (Participants) | 24 | 0 | 11
  Week 32 IGA <=2 n==24,0,11 | 11 |  | 7
  Week 32 IGA improvement. >=2 n==24,0,11: number analyzed (Participants) | 24 | 0 | 11
  Week 32 IGA improvement. >=2 n==24,0,11 | 5 |  | 5
  Week 32 IGA 0/1 n==24,0,11: number analyzed (Participants) | 24 | 0 | 11
  Week 32 IGA 0/1 n==24,0,11 | 4 |  | 4

5. Secondary Outcome: Number (%) of Subjects in Each Category in Physician´s Assessment of Surface Area of Disease (PSAD) - CLP (BOCF) - Entire Treatment Period (FAS)
Description: The Physician Assessment of Surface Area of Disease (PSAD) evaluates the extent of cutaneous lesions estimated by investigator or qualified designee. Assessment scores range from 0-5, with lower scores corresponding to lower percentages of surface area with disease: 0=clear, 1=<2%, 2=2-9%, 3=10-29%, 4=30-50%, 5=>50% of total body surface
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, 28, and 32
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | AIN457 300 mg Q4W - TP 1 and TP 2 - CLP Cohort | Placebo - TP 1 - CLP Cohort | Placebo to AIN457 300 mg Q2W - TP 2 - CLP Cohort
Number analyzed (Participants) | 25 | 12 | 10
Participants
  Baseline 0 Score: number analyzed (Participants) | 25 | 12 | 0
  Baseline 0 Score | 0 | 0 |
  Baseline 1 score: number analyzed (Participants) | 25 | 12 | 0
  Baseline 1 score | 3 | 0 |
  Baseline 2 score: number analyzed (Participants) | 25 | 12 | 0
  Baseline 2 score | 6 | 0 |
  Baseline 3 score: number analyzed (Participants) | 24 | 11 | 0
  Baseline 3 score | 6 | 3 |
  Baseline 4 score: number analyzed (Participants) | 24 | 11 | 0
  Baseline 4 score | 5 | 6 |
  Baseline 5 score: number analyzed (Participants) | 24 | 11 | 0
  Baseline 5 score | 5 | 3 |
  Week 2 0 score: number analyzed (Participants) | 25 | 11 | 0
  Week 2 0 score | 0 | 0 | 0
  Week 2 1 score: number analyzed (Participants) | 25 | 11 | 0
  Week 2 1 score | 6 | 0 |
  Week 2 2 score: number analyzed (Participants) | 25 | 11 | 0
  Week 2 2 score | 5 | 1 |
  Week 2 3 score: number analyzed (Participants) | 25 | 12 | 0
  Week 2 3 score | 9 | 3 |
  Week 2 4 score: number analyzed (Participants) | 25 | 12 | 0
  Week 2 4 score | 3 | 5 |
  Week 2 5 score: number analyzed (Participants) | 25 | 12 | 0
  Week 2 5 score | 2 | 3 |
  Week 4 0 score: number analyzed (Participants) | 25 | 12 | 0
  Week 4 0 score | 0 | 0 |
  Week 4 1 score: number analyzed (Participants) | 25 | 12 | 0
  Week 4 1 score | 3 | 0 |
  Week 4 2 score: number analyzed (Participants) | 25 | 12 | 0
  Week 4 2 score | 8 | 0 |
  Week 4 3 score: number analyzed (Participants) | 25 | 12 | 0
  Week 4 3 score | 8 | 3 |
  Week 4 4 score: number analyzed (Participants) | 25 | 12 | 0
  Week 4 4 score | 3 | 5 |
  Week 4 5 score: number analyzed (Participants) | 25 | 12 | 0
  Week 4 5 score | 2 | 3 |
  Week 8 0 score: number analyzed (Participants) | 25 | 12 | 0
  Week 8 0 score | 0 | 0 |
  Week 8 1 score: number analyzed (Participants) | 25 | 12 | 0
  Week 8 1 score | 7 | 1 |
  Week 8 2 score: number analyzed (Participants) | 25 | 12 | 0
  Week 8 2 score | 5 | 1 |
  Week 8 3 score: number analyzed (Participants) | 24 | 11 | 0
  Week 8 3 score | 7 | 2 |
  Week 8 4 score: number analyzed (Participants) | 24 | 11 | 0
  Week 8 4 score | 4 | 4 |
  Week 8 5 score: number analyzed (Participants) | 24 | 11 | 0
  Week 8 5 score | 2 | 3 |
  Week 12 0 score: number analyzed (Participants) | 25 | 0 | 0
  Week 12 0 score | 0 | 0 |
  Week 12 1 score: number analyzed (Participants) | 25 | 12 | 0
  Week 12 1 score | 6 | 1 |
  Week 12 2 score: number analyzed (Participants) | 25 | 12 | 0
  Week 12 2 score | 7 | 2 |
  Week 12 3 score: number analyzed (Participants) | 23 | 12 | 0
  Week 12 3 score | 7 | 0 |
  Week 12 4 score: number analyzed (Participants) | 23 | 12 | 0
  Week 12 4 score | 3 | 7 |
  Week 12 5 score: number analyzed (Participants) | 23 | 12 | 0
  Week 12 5 score | 2 | 2 |
  Week 16 0 score: number analyzed (Participants) | 24 | 12 | 9
  Week 16 0 score | 0 | 0 | 0
  Week 16 1 score: number analyzed (Participants) | 24 | 12 | 9
  Week 16 1 score | 4 | 2 | 0
  Week 16 2 score: number analyzed (Participants) | 24 | 12 | 9
  Week 16 2 score | 12 | 3 | 3
  Week 16 3 score | 5 | 3 | 3
  Week 16 4 score | 2 | 4 | 4
  Week 16 5 score | 2 | 0 | 0
  Week 20 0 score: number analyzed (Participants) | 25 | 0 | 10
  Week 20 0 score | 0 |  | 0
  Week 20 1 score: number analyzed (Participants) | 25 | 0 | 10
  Week 20 1 score | 6 |  | 0
  Week 20 2 score: number analyzed (Participants) | 25 | 0 | 10
  Week 20 2 score | 12 |  | 3
  Week 20 3 score: number analyzed (Participants) | 25 | 0 | 10
  Week 20 3 score | 3 |  | 2
  Week 20 4 score: number analyzed (Participants) | 25 | 0 | 10
  Week 20 4 score | 1 |  | 3
  Week 20 5 score: number analyzed (Participants) | 25 | 0 | 10
  Week 20 5 score | 2 |  | 2
  Week 24 0 score: number analyzed (Participants) | 25 | 0 | 10
  Week 24 0 score | 1 |  | 0
  Week 24 1 score: number analyzed (Participants) | 25 | 0 | 10
  Week 24 1 score | 8 |  | 0
  Week 24 2 score: number analyzed (Participants) | 25 | 0 | 10
  Week 24 2 score | 10 |  | 2
  Week 24 3 score: number analyzed (Participants) | 25 | 0 | 10
  Week 24 3 score | 1 |  | 2
  Week 24 4 score: number analyzed (Participants) | 25 | 0 | 10
  Week 24 4 score | 2 |  | 4
  Week 24 5 score: number analyzed (Participants) | 25 | 0 | 10
  Week 24 5 score | 3 |  | 2
  Week 28 0 score: number analyzed (Participants) | 25 | 0 | 10
  Week 28 0 score | 0 |  | 0
  Week 28 1 score: number analyzed (Participants) | 25 | 0 | 10
  Week 28 1 score | 6 |  | 0
  Week 28 2 score: number analyzed (Participants) | 25 | 0 | 10
  Week 28 2 score | 11 |  | 2
  Week 28 3 score: number analyzed (Participants) | 25 | 0 | 10
  Week 28 3 score | 1 |  | 3
  Week 28 4 score: number analyzed (Participants) | 25 | 0 | 10
  Week 28 4 score | 3 |  | 3
  Week 28 5 score: number analyzed (Participants) | 25 | 0 | 10
  Week 28 5 score | 2 |  | 2
  Week 32 0 score: number analyzed (Participants) | 25 | 0 | 10
  Week 32 0 score | 2 |  | 0
  Week 32 1 score: number analyzed (Participants) | 25 | 0 | 10
  Week 32 1 score | 5 |  | 1
  Week 32 2 score: number analyzed (Participants) | 25 | 0 | 10
  Week 32 2 score | 10 |  | 0
  Week 32 3 score: number analyzed (Participants) | 25 | 0 | 10
  Week 32 3 score | 3 |  | 4
  Week 32 4 score: number analyzed (Participants) | 25 | 0 | 10
  Week 32 4 score | 1 |  | 2
  Week 32 5 score: number analyzed (Participants) | 25 | 0 | 10
  Week 32 5 score | 3 |  | 2

6. Secondary Outcome: Number (%) of Subjects With Dermatology Life Quality Index Response Scores of 0 to 1 up to Week 32 - CLP Cohort - Entire Treatment Period (FAS)
Description: The Dermatology Life Quality Index (DLQI) is a 10-item general dermatology disability index designed to assess health-related quality of life (HRQoL) in adult subjects with skin diseases such as eczema, psoriasis, acne, and viral warts. The measure is self-administered and includes domains of daily activities, leisure, personal relationships, symptoms and feelings, treatment, and work/school. The recall period is the last week, and the instrument requires 1 to 2 minutes for completion. Each item has four response categories ranging from 0 (not at all) to 3 (very much). "Not relevant" is also a valid response and is scored as 0. The DLQI total score is a sum of the 10 questions. Scores range from 0 to 30, with higher scores indicating greater HRQoL impairment.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, and 32
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | AIN457 300 mg Q4W - TP 1 and TP 2 - CLP Cohort | Placebo - TP 1 - CLP Cohort | Placebo to AIN457 300 mg Q2W - TP 2 - CLP Cohort
Number analyzed (Participants) | 25 | 12 | 10
Participants
  Baseline n=25,12,0: number analyzed (Participants) | 25 | 12 | 0
  Baseline n=25,12,0 | 0 | 0 |
  Week 4 n=24,11,0: number analyzed (Participants) | 24 | 11 | 0
  Week 4 n=24,11,0 | 2 | 0 |
  Week 8 n=25,11,0: number analyzed (Participants) | 25 | 11 | 0
  Week 8 n=25,11,0 | 2 | 0 |
  Week 12 n=25,12,0: number analyzed (Participants) | 25 | 12 | 0
  Week 12 n=25,12,0 | 3 | 1 |
  Week 16 n=25,12,10 | 3 | 2 | 2
  Week 20 n=24,0,10: number analyzed (Participants) | 24 | 0 | 10
  Week 20 n=24,0,10 | 3 |  | 1
  Week 24 n=25,0,10: number analyzed (Participants) | 25 | 0 | 10
  Week 24 n=25,0,10 | 4 |  | 1
  Week 28 n=23,0,10: number analyzed (Participants) | 23 | 0 | 10
  Week 28 n=23,0,10 | 3 |  | 1
  Week 32 n=25,0,9: number analyzed (Participants) | 25 | 0 | 9
  Week 32 n=25,0,9 | 2 |  | 1

7. Secondary Outcome: Number (%) of Subjects With Dermatology Life Quality Index Response Scores of 0 to 1 up to Week 32 - MLP Cohort - Entire Treatment Period (FAS)
Description: The DLQI is a 10-item general dermatology disability index designed to assess health-related quality of life (HRQoL) in adult subjects with skin diseases such as eczema, psoriasis, acne, and viral warts (Finlay and Khan 1994). The measure is self-administered and includes domains of daily activities, leisure, personal relationships, symptoms and feelings, treatment, and work/school. The recall period is the last week, and the instrument requires 1 to 2 minutes for completion. Each item has four response categories ranging from 0 (not at all) to 3 (very much). "Not relevant" is also a valid response and is scored as 0. The DLQI total score is a sum of the 10 questions. Scores range from 0 to 30, with higher scores indicating greater HRQoL impairment.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, and 32
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- AIN457 300 mg Q4W - TP 1 and TP 2- MLP Cohort: AIN457 300 mg every 4 weeks administered via a pre-filled syringe. Participants on AIN457 in TP 1 for 16 weeks continued AIN457 in TP 2 for 16 weeks.
Arm/Group | AIN457 300 mg Q4W - TP 1 and TP 2- MLP Cohort | Placebo - TP 1 - MLP Cohort | Placebo to AIN457 300 mg Q2W TP 2 - MLP Cohort
Number analyzed (Participants) | 24 | 13 | 11
Participants
  Baseline n=24,13,0: number analyzed (Participants) | 24 | 13 | 0
  Baseline n=24,13,0 | 0 | 0 |
  Week 4 n=24,13,0: number analyzed (Participants) | 24 | 13 | 0
  Week 4 n=24,13,0 | 2 | 1 |
  Week 8 n=24,13,0: number analyzed (Participants) | 24 | 13 | 0
  Week 8 n=24,13,0 | 4 | 1 |
  Week 12 n=24,13,0: number analyzed (Participants) | 24 | 13 | 0
  Week 12 n=24,13,0 | 4 | 2 |
  Week 16 n=24,13,11 | 5 | 3 | 2
  Week 20 n=24,0,11: number analyzed (Participants) | 24 | 0 | 11
  Week 20 n=24,0,11 | 7 |  | 2
  Week 24 n=24,0,10: number analyzed (Participants) | 24 | 0 | 10
  Week 24 n=24,0,10 | 7 |  | 3
  Week 28 n=23,0,11: number analyzed (Participants) | 23 | 0 | 11
  Week 28 n=23,0,11 | 3 |  | 2
  Week 32 n=23,0,10: number analyzed (Participants) | 23 | 0 | 10
  Week 32 n=23,0,10 | 4 |  | 2

8. Secondary Outcome: Number (%) of Subjects With Dermatology Life Quality Index Response Scores of 0 to 1 up to Week 32 - LPP Cohort - Entire Treatment Period (FAS)
Description: as for outcome 7
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, and 32
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Placebo to AIN457 300 mg Q2W TP 2 - LPP Cohort: Placebo non-responders during TP 1 received AIN457 300 mg every 2 weeks from Week 16 to Week 32 in TP 2 via a pre-filled syringe.
Arm/Group | AIN457 300 mg Q4W - TP 1 and TP 2 - LPP Cohort | Placebo - TP 1 - LPP Cohort | Placebo to AIN457 300 mg Q2W TP 2 - LPP Cohort
Number analyzed (Participants) | 24 | 13 | 13
Participants
  Baseline n=24,13,0: number analyzed (Participants) | 24 | 13 | 0
  Baseline n=24,13,0 | 0 | 0 |
  Week 4 n=24,13,0: number analyzed (Participants) | 24 | 13 | 0
  Week 4 n=24,13,0 | 3 | 1 |
  Week 8 n=24,13,0: number analyzed (Participants) | 24 | 13 | 0
  Week 8 n=24,13,0 | 3 | 1 |
  Week 12 n=24,13,0: number analyzed (Participants) | 24 | 13 | 0
  Week 12 n=24,13,0 | 2 | 2 |
  Week 16 n=24,13,13 | 2 | 1 | 1
  Week 20 n=24,0,13: number analyzed (Participants) | 24 | 0 | 13
  Week 20 n=24,0,13 | 4 |  | 3
  Week 24 n=23,0,13: number analyzed (Participants) | 23 | 0 | 13
  Week 24 n=23,0,13 | 2 |  | 3
  Week 28 n=24,0,13: number analyzed (Participants) | 24 | 0 | 13
  Week 28 n=24,0,13 | 2 |  | 2
  Week 32 n=24,0,11: number analyzed (Participants) | 24 | 0 | 11
  Week 32 n=24,0,11 | 1 |  | 3

9. Secondary Outcome: Summary of Baseline Score and Change From Baseline for Patient Assessment of Itch Using Numeric Rating Scale (NRS) by Question - CLP Cohort (BOCF) (FAS)
Description: Itch is assessed with the following questions: • "Overall, how severe was your lichen planus-related itching during the past 24 hours?" • "How severe was your lichen planus-related itching at the worst moment during the past 24 hours?" • "Overall, how bothered were you by your lichen planus-related itching during the past 24 hours?" Answers are given on a numeric rating scale (NRS) from 0 to 10, with 0 meaning "no itch" and 10 meaning "the worst itch imaginable".
Time Frame: Baseline, Week 16 and Week 32
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Placebo to AIN457 300 mg Q2W TP 2 - CLP Cohort: Placebo non-responders during TP 1 received AIN457 300 mg every 2 weeks up to 16 weeks administered via a pre-filled syringe.
Arm/Group | AIN457 300 mg Q4W - TP 1 and TP 2 - CLP Cohort | Placebo - TP 1 - CLP Cohort | Placebo to AIN457 300 mg Q2W TP 2 - CLP Cohort
Number analyzed (Participants) | 25 | 12 | 10
scores on a scale
  Baseline - Question 1 | 5.1 (2.66) | 5.7 (2.77) | 5.8 (3.01)
  Week 16 Severity of itch during past 24 hours n=25,12,10 | -0.8 (1.91) | -2.3 (3.25) | -2.0 (3.53)
  Week 32 Severity of itch during past 24 hours n=25,0,9: number analyzed (Participants) | 25 | 0 | 9
  Week 32 Severity of itch during past 24 hours n=25,0,9 | -1.5 (2.24) |  | -1.1 (2.42)
  Baseline- Question 2 | 5.6 (2.72) | 6.3 (2.86) | 5.9 (3.03)
  Week 16 How severe was itch at worst moment during past 24 hours n=25,12,10 | -0.9 (2.52) | -2.7 (3.73) | -1.9 (3.54)
  Week 32 How severe was itch at worst moment during past 24 hours n=25,0,9: number analyzed (Participants) | 25 | 0 | 9
  Week 32 How severe was itch at worst moment during past 24 hours n=25,0,9 | -1.3 (2.13) |  | -1.2 (2.49)
  Baseline- Question 3 | 4.8 (3.08) | 6.1 (2.94) | 6.1 (3.21)
  Week 16 How bothered by Itch during past 24 hours n=25,12,10 | -1.0 (2.65) | -2.7 (3.55) | -2.4 (3.84)
  Week 32 How bothered by Itch during past 24 hours n=25,0,9: number analyzed (Participants) | 25 | 0 | 9
  Week 32 How bothered by Itch during past 24 hours n=25,0,9 | -1.1 (2.45) |  | -1.2 (2.28)

10. Secondary Outcome: Summary of Baseline Score and Change From Baseline for Patient Assessment of Itch Using Numeric Rating Scale (NRS) by Question - MLP Cohort (BOCF) (FAS)
Description: as for outcome 9
Time Frame: Baseline, Week 16 and Week 32
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | AIN457 300 mg Q4W - TP 1 and TP 2 - MLP Cohort | Placebo - TP 1 - MLP Cohort | Placebo to AIN457 300 mg Q2W TP 2 - MLP Cohort
Number analyzed (Participants) | 24 | 13 | 11
scores on a scale
  Baseline - Question 1 n=23,13,11: number analyzed (Participants) | 23 | 13 | 11
  Baseline - Question 1 n=23,13,11 | 2.5 (2.83) | 3.8 (3.81) | 4.3 (3.93)
  Week 16 Severity of itch during past 24 hours n=23,13,11: number analyzed (Participants) | 23 | 13 | 11
  Week 16 Severity of itch during past 24 hours n=23,13,11 | 0.3 (3.26) | -0.2 (3.41) | -0.3 (3.72)
  Week 32 Severity of itch during past 24 hours n=22,0,10: number analyzed (Participants) | 22 | 0 | 10
  Week 32 Severity of itch during past 24 hours n=22,0,10 | 0.1 (2.97) |  | -0.4 (3.37)
  Baseline - Question 2 n=23,13,11: number analyzed (Participants) | 23 | 13 | 11
  Baseline - Question 2 n=23,13,11 | 2.4 (2.90) | 3.6 (3.99) | 4.1 (4.16)
  Week 16 How severe was itch at worst moment during past 24 hours n=23,13,11: number analyzed (Participants) | 23 | 13 | 11
  Week 16 How severe was itch at worst moment during past 24 hours n=23,13,11 | 0.8 (3.04) | 0.4 (3.25) | 0.4 (3.56)
  Week 32 How severe was itch at worst moment during past 24 hours n=22,0,10: number analyzed (Participants) | 22 | 0 | 10
  Week 32 How severe was itch at worst moment during past 24 hours n=22,0,10 | 0.3 (2.43) |  | 0.4 (3.81)
  Baseline - Question 3 n=24,13,11 | 3.4 (3.41) | 4.0 (4.14) | 4.5 (4.27)
  Week 16 How bothered by Itch during past 24 hours n=23,13,11: number analyzed (Participants) | 23 | 13 | 11
  Week 16 How bothered by Itch during past 24 hours n=23,13,11 | -0.5 (2.95) | 0.1 (3.12) | 0.0 (3.41)
  Week 32 How bothered by Itch during past 24 hours n=22,0,10: number analyzed (Participants) | 22 | 0 | 10
  Week 32 How bothered by Itch during past 24 hours n=22,0,10 | -0.2 (1.33) |  | -0.4 (4.25)

11. Secondary Outcome: Summary of Baseline Score and Change From Baseline for Patient Assessment of Itch Using Numeric Rating Scale (NRS) by Question - LPP Cohort (BOCF) (FAS)
Description: as for outcome 9
Time Frame: Baseline, Week 16 and Week 32
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Placebo to AIN457 300 mg Q2W - TP 2 - LPP Cohort: Placebo non-responders during TP 1 received AIN457 300 mg every 2 weeks from Week 16 to Week 32 in TP 2 via a pre-filled syringe.
Arm/Group | AIN457 300 mg Q4W - TP 1 and TP 2 - LPP Cohort | Placebo - TP 1 - LPP Cohort | Placebo to AIN457 300 mg Q2W - TP 2 - LPP Cohort
Number analyzed (Participants) | 24 | 13 | 13
scores on a scale
  Baseline - Question 1 n=24,13,13 | 4.5 (2.25) | 3.8 (2.68) | 3.8 (2.68)
  Week 16 Severity of itch during past 24 hours n=24,13,11: number analyzed (Participants) | 24 | 13 | 11
  Week 16 Severity of itch during past 24 hours n=24,13,11 | -0.5 (2.25) | -1.1 (2.47) | -1.1 (2.47)
  Week 32 Severity of itch during past 24 hours n=24,0,11: number analyzed (Participants) | 24 | 0 | 11
  Week 32 Severity of itch during past 24 hours n=24,0,11 | -1.6 (2.06) |  | -2.4 (2.84)
  Baseline - Question 2 n=24,13,13 | 5.1 (2.43) | 4.2 (2.86) | 4.1 (4.16)
  Week 16 How severe was itch at worst moment during past 24 hours n=24,13,13 | -0.7 (2.35) | -1.3 (2.81) | -1.3 (2.81)
  Week 32 How severe was itch at worst moment during past 24 hours n=24,0,11: number analyzed (Participants) | 24 | 0 | 11
  Week 32 How severe was itch at worst moment during past 24 hours n=24,0,11 | -1.8 (2.23) |  | -2.6 (3.01)
  Baseline - Question 3 n=24,13,11: number analyzed (Participants) | 24 | 13 | 11
  Baseline - Question 3 n=24,13,11 | 4.0 (2.36) | 3.2 (2.79) | 3.2 (2.79)
  Week 16 How bothered by Itch during past 24 hours n=24,13,13 | -0.4 (2.43) | -1.2 (3.02) | -1.2 (3.02)
  Week 32 How bothered by Itch during past 24 hours n=24,0,11: number analyzed (Participants) | 24 | 0 | 11
  Week 32 How bothered by Itch during past 24 hours n=24,0,11 | -1.7 (2.08) |  | -2.2 (2.44)

12. Secondary Outcome: Summary of Baseline Score and Change From Baseline for Patient Assessment of Pain Using Numeric Rating Scale (NRS) by Question - CLP Cohort (BOCF) (FAS)
Description: Pain is assessed with the following questions: • "Overall, how severe was your lichen planus-related pain during the past 24 hours?" • "How severe was your lichen planus-related pain at the worst moment during the past 24 hours?" • "Overall, how bothered were you by your lichen planus-related pain during the past 24 hours?" Answers are given on a numeric rating scale (NRS) from 0 to 10, with 0 meaning "no pain" and 10 meaning "the worst pain imaginable".
Time Frame: Baseline, Week 16 and Week 32
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | AIN457 300 mg Q4W - TP 1 and TP 2 - CLP Cohort | Placebo - TP 1 - CLP Cohort | Placebo to AIN457 300 mg Q2W - TP 2 - CLP Cohort
Number analyzed (Participants) | 25 | 12 | 10
scores on a scale
  Baseline - Question 1 n=25,12,10 | 1.09 (2.05) | 3.4 (2.61) | 3.5 (2.51)
  Week 16 Severity of pain during past 24 hours n=25,12,10 | 0.2 (1.48) | -0.8 (1.40) | -0.8 (1.48)
  Week 32 Severity of pain during past 24 hours n=25,0,9: number analyzed (Participants) | 25 | 0 | 9
  Week 32 Severity of pain during past 24 hours n=25,0,9 | -0.3 (1.65) |  | -0.3 (2.29)
  Baseline - Question 2 n=25,12,10 | 2.2 (2.48) | 3.9 (3.23) | 3.9 (3.03)
  Week 16 How severe was pain at worst moment during past 24 hours n=25,12,10 | 0.1 (2.03) | -1.2 (1.70) | -1.0 (1.56)
  Week 32 How severe was pain at worst moment during past 24 hours n=25,0,9: number analyzed (Participants) | 25 | 0 | 9
  Week 32 How severe was pain at worst moment during past 24 hours n=25,0,9 | -0.4 (2.35) |  | -0.4 (2.70)
  Baseline - Question 3 n=25,12,10 | 2.1 (2.55) | 3.7 (2.96) | 3.8 (2.94)
  Week 16 How bothered by pain during past 24 hour n=25,12,10 | 0.1 (2.09) | -0.6 (1.62) | 0.5 (1.72)
  Week 32 How bothered by pain during past 24 hours n=25, 0,9: number analyzed (Participants) | 25 | 0 | 9
  Week 32 How bothered by pain during past 24 hours n=25, 0,9 | -0.2 (1.71) |  | -0.3 (2.45)

13. Secondary Outcome: Summary of Baseline Score and Change From Baseline for Patient Assessment of Pain Using Numeric Rating Scale (NRS) by Question -MLP Cohort (BOCF) (FAS)
Description: as for outcome 12
Time Frame: Baseline, Week 16 and Week 32
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | AIN457 300 mg Q4W - TP 1 and TP 2 - MLP Cohort | Placebo - TP 1 - MLP Cohort | Placebo to AIN457 300 mg Q2W TP 2 - MLP Cohort
Number analyzed (Participants) | 24 | 13 | 11
scores on a scale
  Baseline - Question 1 n=24,13,11 | 5.1 (2.86) | 5.9 (3.09) | 6.3 (3.23)
  Week 16 Severity of pain during past 24 hours n=24,13,11 | -0.5 (3.08) | -0.1 (3.01) | 0.0 (3.29)
  Week 32 Severity of pain during past 24 hours n=23,0,10: number analyzed (Participants) | 23 | 0 | 10
  Week 32 Severity of pain during past 24 hours n=23,0,10 | -0.3 (2.18) |  | -0.6 (2.59)
  Baseline - Question 2 n=24,13,11 | 5.4 (2.99) | 6.4 (3.15) | 6.7 (3.26)
  Week 16 How severe was pain at worst moment during past 24 hours n=24,13,11 | -0.5 (3.13) | -0.3 (2.75) | -0.2 (2.99)
  Week 32 How severe was pain at worst moment during past 24 hours n=23,0,10: number analyzed (Participants) | 23 | 0 | 10
  Week 32 How severe was pain at worst moment during past 24 hours n=23,0,10 | -0.3 (2.06) |  | -0.5 (2.46)
  Baseline - Question 3 n=24,13,11 | 5.5 (3.35) | 6.5 (2.76) | 6.8 (2.79)
  Week 16 How bothered by pain during past 24 hour n=24,13,11 | -0.8 (3.54) | -0.3 (2.21) | -0.1 (2.34)
  Week 32 How bothered by pain during past 24 hours n=23,0,10: number analyzed (Participants) | 23 | 0 | 10
  Week 32 How bothered by pain during past 24 hours n=23,0,10 | -0.5 (2.74) |  | -0.9 (2.69)

14. Secondary Outcome: Summary of Baseline Score and Change From Baseline for Patient Assessment of Pain Using Numeric Rating Scale (NRS) by Question - LPP Cohort (BOCF) (FAS)
Description: as for outcome 12
Time Frame: Baseline, Week 16 and Week 32
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | AIN457 300 mg Q4W - TP 1 and TP 2 - LPP Cohort | Placebo - TP 1 - LPP Cohort | Placebo to AIN457 300 mg Q2W - TP 2 - LPP Cohort
Number analyzed (Participants) | 24 | 13 | 12
scores on a scale
  Baseline - Question 1 n=24,13,12 | 2.5 (2.43) | 2.0 (2.38) | 2.0 (2.38)
  Week 16 Severity of pain during past 24 hours n=24,13,12 | 0.3 (2.61) | -0.5 (1.90) | -0.5 (1.90)
  Week 32 Severity of pain during past 24 hours n=24,0,11: number analyzed (Participants) | 24 | 0 | 11
  Week 32 Severity of pain during past 24 hours n=24,0,11 | -0.6 (1.72) |  | -1.5 (2.02)
  Baseline - Question 2 24,13,12 | 2.8 (2.68) | 2.5 (2.73) | 2.5 (2.73)
  Week 16 How severe was pain at worst moment during past 24 hours n=24,13,12 | 0.2 (3.16) | -0.9 (2.25) | -0.9 (2.25)
  Week 32 How severe was pain at worst moment during past 24 hours n=24,0,11: number analyzed (Participants) | 24 | 0 | 11
  Week 32 How severe was pain at worst moment during past 24 hours n=24,0,11 | -0.8 (2.06) |  | -2.0 (2.45)
  Baseline - Question 3 n=24,13,12 | 2.7 (2.56) | 2.4 (2.75) | 2.4 (2.75)
  Week 16 How bothered by pain during past 24 hour n=24,13,12 | 0.0 (2.87) | -1.1 (2.25) | -1.1 (2.25)
  Week 32 How bothered by pain during past 24 hours n=24,0,11: number analyzed (Participants) | 24 | 0 | 11
  Week 32 How bothered by pain during past 24 hours n=24,0,11 | -0.8 (1.79) |  | -1.9 (2.51)

15. Secondary Outcome: Summary of Baseline Score and Change From Baseline in Reticular Erythematous Ulcerative Score (REU) - MLP Cohort - (BOCF) - Entire Treatment Period
Description: REU measured disease severity based on 3 dimensions: reticulation, erythema and ulceration for all subjects in the MLP cohort who had an oral presentation of the disease. The total score ranged from 0-115 with higher values corresponding to higher activity of the disease.
Time Frame: Baseline, Week 16 and Week 32
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | AIN457 300 mg Q4W - TP 1 and TP 2 - MLP Cohort | Placebo - TP 1 - MLP Cohort | Placebo to AIN457 300 mg Q2W TP 2 - MLP Cohort
Number analyzed (Participants) | 21 | 13 | 10
scores on a scale
  Baseline n=21,12,10: number analyzed (Participants) | 21 | 12 | 10
  Baseline n=21,12,10 | 21.31 (8.747) | 25.29 (9.102) | 26.95 (8.855)
  Week 16 n=21,12,10: number analyzed (Participants) | 21 | 12 | 10
  Week 16 n=21,12,10 | -4.83 (11.102) | -5.79 (14.476) | -4.10 (15.196)
  Week 32 n=20,0,9: number analyzed (Participants) | 20 | 0 | 9
  Week 32 n=20,0,9 | -6.08 (10.206) |  | -2.17 (15.802)

16. Secondary Outcome: Summary of Baseline Score and Change From Baseline in Oral Lichen Planus Symptom Severity Measure (OLPSSM) - MLP Cohort - (BOCF) - Entire Treatment Period
Description: OLPSSM is a self-administered assessment of the symptom experience of subjects with oral LP in clinical studies. It includes 7 triggers contributing to soreness of oral lichen planus: Brushing teeth, eating food, drinking liquids, smiling, breathing through mouth, talking and touching. These 7 items contributed equally to a total OLP symptom severity score, ranging from 0 to 28, with higher scores indicating worse severity.
Time Frame: Baseline, Week 16 and Week 32
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | AIN457 300 mg Q4W - TP 1 and TP 2 - MLP Cohort | Placebo - TP 1 - MLP Cohort | Placebo to AIN457 300 mg Q2W TP 2 - MLP Cohort
Number analyzed (Participants) | 21 | 12 | 10
scores on a scale
  Baseline n=21,12,10 | 11.0 (5.98) | 13.4 (5.50) | 13.9 (5.78)
  Week 16 n=21,12,10 | -1.0 (6.82) | 0.8 (6.47) | -0.4 (7.09)
  Week 32 n=20,0,9: number analyzed (Participants) | 20 | 0 | 9
  Week 32 n=20,0,9 | -1.8 (5.67) |  | -0.7 (7.00)

17. Secondary Outcome: Summary of Baseline Score and Change From Baseline for Lichen Planopilaris Activity Index (LPPAI)- LPP Cohort (BOCF) (FAS)
Description: The LPPAI assesses symptoms (pruritus, pain, burning), signs (erythema, perifollicular erythema and scale), a measure of activity (pull test) and extension of disease. These subjective and objective measures are assigned numeric values to establish a disease activity score. The total score ranges from 0 to 10, with higher scores corresponding to higher disease activity
Time Frame: Baseline, Week 16 and Week 32
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | AIN457 300 mg Q4W - TP 1 and TP 2 - LPP Cohort | Placebo - TP 1 - LPP Cohort | Placebo to AIN457 300 mg Q2W TP 2 - Lpp Cohort
Number analyzed (Participants) | 24 | 13 | 13
scores on a scale
  Baseline n=24,13,13 | 5.92 (2.071) | 5.95 (1.767) | 5.95 (1.767)
  Week 16 n=24,13,13 | -1.44 (2.517) | -2.24 (2.522) | -2.24 (2.522)
  Week 32 n=24,0,13: number analyzed (Participants) | 24 | 0 | 13
  Week 32 n=24,0,13 | -2.44 (2.428) |  | -3.20 (2.927)

18. Secondary Outcome: Summary of Baseline Score and Change From Baseline for Scalpdex - LPP Cohort (BOCF) (FAS)
Description: Scalpdex is a self-administered, health-related quality of life instrument originally developed for scalp dermatitis. This survey includes 23 items, each item scored on a scale of 0-100, where 0=never, 25=rarely, 50=sometimes, 75=often and 100=all the time. The 23 items pertain to 3 domains: symptom, emotions and functioning. Subjects were asked to score themselves on how true each of the 23 statements has been for them over the past four weeks. the total score is the average of the scores of the 23 items. A higher total score indicated a higher impairment in quality of life.
Time Frame: Baseline, Week 16 and Week 32
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- AIN457 300 mg Q4W - TP 1 and TP 2 -LPP Cohort: AIN457 300 mg every 4 weeks administered via a pre-filled syringe. Participants on AIN457 in TP 1 for 16 weeks continued AIN457 in TP 2 for 16 weeks.
Arm/Group | AIN457 300 mg Q4W - TP 1 and TP 2 -LPP Cohort | Placebo - TP 1 - LPP Cohort | Placebo to AIN457 300 mg Q2W - TP 2 - LPP Cohort
Number analyzed (Participants) | 24 | 13 | 12
scores on a scale
  Baseline n=24,13,12 | 55.75 (16.476) | 54.01 (23.252) | 54.01 (23.252)
  Week 16 n=24,13,12 | 1.86 (10.695) | -6.94 (11.508) | -6.94 (11.508)
  Week 32 n=24,0,11: number analyzed (Participants) | 24 | 0 | 11
  Week 32 n=24,0,11 | -4.26 (12.876) |  | -14.43 (16.464)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment up to a maximum of 300 days which included an approximate follow up period of 8 weeks for AIN457 treatment groups.
Description: "Any AIN457 300 mg Q4W" Arm/Group Total Number at Risk represents all participants who were assigned AIN457 300 mg Q4W for a given cohort during the study. Participants who were on placebo in Treatment Period 1 who continued into Treatment Period 2 received AIN457 300 mg Q2W.
Groups:
- AIN457 300 mg Q4W - CLP Cohort; AIN457 300 mg Q4W - MLP Cohort: AIN457 300 mg every 4 weeks up to 32 weeks administered via a pre-filled syringe
- Placebo - CLP Cohort; Placebo - MLP Cohort; Placebo - LPP Cohort: Matching placebo administered every 4 weeks up to 16 weeks via a pre-filled syringe
- Any AIN457 300 mg - CLP Cohort; Any AIN457 300 mg - MLP Cohort; Any AIN457 300 mg - LPP Cohort: AIN457 300mg administered every 4 weeks or every 2 weeks via a pre-filled syringe
- Placebo to AIN457 300 mg Q2W - CLP Cohort; Placebo to AIN457 300 mg Q2W - MLP Cohort; Placebo to AIN457 300 mg Q2W - LPP Cohort: Placebo non-responders during TP 1 received AIN457 300 mg every 2 weeks from Week 16 to Week 32 in TP 2 via a pre-filled syringe.
- AIN457 300 mg Q4W - LPP Cohort: AIN457457 300 mg every 4 weeks up to 32 weeks administered via a pre-filled syringe
Arm/Group | AIN457 300 mg Q4W - CLP Cohort | Placebo - CLP Cohort | Any AIN457 300 mg - CLP Cohort | Placebo to AIN457 300 mg Q2W - CLP Cohort | AIN457 300 mg Q4W - MLP Cohort | Placebo - MLP Cohort | Any AIN457 300 mg - MLP Cohort | Placebo to AIN457 300 mg Q2W - MLP Cohort | AIN457 300 mg Q4W - LPP Cohort | Placebo - LPP Cohort | Any AIN457 300 mg - LPP Cohort | Placebo to AIN457 300 mg Q2W - LPP Cohort
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/12 | 0/33 | 0/8 | 0/24 | 0/13 | 0/35 | 0/11 | 0/24 | 0/13 | 0/36 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/25 | 1/12 | 0/33 | 0/8 | 1/24 | 0/13 | 2/35 | 1/11 | 0/24 | 1/13 | 1/36 | 1/12
Other Adverse Events (participants affected / at risk) | 15/25 | 7/12 | 21/33 | 6/8 | 18/24 | 8/13 | 26/35 | 8/11 | 16/24 | 7/13 | 22/36 | 6/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 300 mg Q4W - CLP Cohort (N=25) | Placebo - CLP Cohort (N=12) | Any AIN457 300 mg - CLP Cohort (N=33) | Placebo to AIN457 300 mg Q2W - CLP Cohort (N=8) | AIN457 300 mg Q4W - MLP Cohort (N=24) | Placebo - MLP Cohort (N=13) | Any AIN457 300 mg - MLP Cohort (N=35) | Placebo to AIN457 300 mg Q2W - MLP Cohort (N=11) | AIN457 300 mg Q4W - LPP Cohort (N=24) | Placebo - LPP Cohort (N=13) | Any AIN457 300 mg - LPP Cohort (N=36) | Placebo to AIN457 300 mg Q2W - LPP Cohort (N=12)
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 300 mg Q4W - CLP Cohort (N=25) | Placebo - CLP Cohort (N=12) | Any AIN457 300 mg - CLP Cohort (N=33) | Placebo to AIN457 300 mg Q2W - CLP Cohort (N=8) | AIN457 300 mg Q4W - MLP Cohort (N=24) | Placebo - MLP Cohort (N=13) | Any AIN457 300 mg - MLP Cohort (N=35) | Placebo to AIN457 300 mg Q2W - MLP Cohort (N=11) | AIN457 300 mg Q4W - LPP Cohort (N=24) | Placebo - LPP Cohort (N=13) | Any AIN457 300 mg - LPP Cohort (N=36) | Placebo to AIN457 300 mg Q2W - LPP Cohort (N=12)
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Auricular swelling (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 2 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 3 | 1 | 1 | 0 | 3 | 2 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukoplakia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0
Injection site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0
Immunisation reaction (Immune system disorders) | 3 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 2 | 1 | 2 | 0 | 4 | 2 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Helicobacter infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes ophthalmic (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 2 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 3 | 1
Oral herpes (Infections and infestations) | 1 | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Post-acute COVID-19 syndrome (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Superinfection (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 1 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Headache (Nervous system disorders) | 3 | 0 | 3 | 0 | 0 | 1 | 2 | 2 | 5 | 2 | 5 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Micturition disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Breast cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Lichen planus (Skin and subcutaneous tissue disorders) | 3 | 1 | 4 | 1 | 4 | 0 | 5 | 1 | 1 | 0 | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 3 | 0 | 3 | 0 | 3 | 1 | 3 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0
Hypertension (Vascular disorders) | 2 | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-10-26): https://cdn.clinicaltrials.gov/large-docs/96/NCT04300296/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-19): https://cdn.clinicaltrials.gov/large-docs/96/NCT04300296/SAP_001.pdf